CLINICAL TRIAL: NCT02806349
Title: Effect of Co-administration of a Konjac-Glucomannan Fibre Blend and American Ginseng (Panax Quinquefolius L.) on Glycemia and Serum Lipids in Well-controlled Type 2 Diabetes: A Randomized Controlled, Clinical Trial
Brief Title: Konjac-Glucomannan Fibre Blend and American Ginseng in Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vladimir Vuksan (Other)
Collaborators: Canadian Diabetes Association (Other)
Responsible Party: Sponsor-Investigator, Vladimir Vuksan, Senior Scientist, Unity Health Toronto
Organization: Unity Health Toronto (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RB02-014C
Record Dates: First submitted 2016-03-02; First posted 2016-06-20 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: American ginseng; Konjac glucomannan fiber
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Asian ginseng

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): 3g/d Cornstarch and 14g/d wheat bran control
  Interventions: Dietary Supplement: Control
- K-GB&AG (Experimental): 3g/d American Ginseng and 7g/d Konjac-glucomannan fiber blend
  Interventions: Dietary Supplement: American Ginseng; Dietary Supplement: Konjac-glucomannan fiber blend

INTERVENTIONS:
Dietary Supplement: American Ginseng — herb
  Other Names: Panax quinquefolius L.
  Arms: K-GB&AG
Dietary Supplement: Konjac-glucomannan fiber blend — Blend of 2 viscous fibers: konjac mannan and xanthan
  Arms: K-GB&AG
Dietary Supplement: Control — Fiber matched control for intervention (corn starch and wheat bran)
  Arms: Control

SUMMARY:
The purpose of this study was to determine whether the co-administration of a konjac-glucomannan fibre blend and American ginseng in a randomized, placebo-controlled, cross-over trial can improve diabetes management.

DETAILED DESCRIPTION:
The study used a partially blinded, randomized, placebo controlled, crossover design. Due to the nature of the fibres it was not possible to blind the participant with respect to type of fibre. The study was divided into two phases with each phase having a four 4-week run-in period, and a 12-week treatment period, separated by a minimum 4-week wash-out period.

The treatments consisted of an ad libitum Canadian Diabetes Association recommended diet supplemented with capsules which contained either cornstarch (control) or AG (test) and a fiber supplement consisting of either wheat bran (control) or a viscous fiber blend of konjac mannan and xanthan (test). Participants were asked to attend the clinic at weeks -4, 0, 3, 6, and 12 during each phase.

Outcome measures There were three levels of outcome measures including efficacy, safety, and compliance. Statistical analysis The results are presented as mean ± SEM and considered statistically significant at p<0.05. Statistical analysis was performed using the SAS version 8.2 (SAS Institute, Cary, NC). Parametric analyses were conducted following a comparison of the sampling distribution to a normal distribution (Shapiro-Wilk and Kolmogorov-Smirnov tests). GLM was used to perform two-way ANOVA to detect differences of outcome variables in treatments and visits, controlling for treatment sequence and sex. If the effect of treatment was significant then percent differences were calculated between weeks 12 of test and control and analyzed using the GLM repeated measures one-way ANOVA controlling for sex. Parametric analyses were conducted following a comparison of the sampling distribution to a normal distribution (Shapiro-Wilk and Kolmogorov-Smirnov tests). The tests did not reject the null hypothesis at α=0.05. All comparisons were paired, thus each participant served as his/her own control. As this was a cross-over study, only participants who completed the study were included in the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes of at least 1 year
* age between 40 and 75 years old
* treated with diet and anti hyperglycemic medications
* HbA1c between 6.5% and 8.4%
* Systolic blood pressure <140mmHg
* Diastolic blood pressure <90mmHg
* Clinically euthyroid
* Normal renal and liver function

Exclusion Criteria:

* treated with insulin
* age less than 40 or older than 75 years old at the start of the trial

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2002-03; Primary Completion 2004-11 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
HbA1c | Week 12
  Difference at week 12 between control and test intervention

SECONDARY OUTCOMES:
Total Cholesterol | Week 12
  Difference at week 12 between control and test intervention
High sensitivity C reactive protein | Week 12
  Difference at week 12 between control and test intervention
Apolipoprotein A and B | Week 12
  Difference at week 12 between control and test intervention
Oxidized LDL | Week 12
  Difference at week 12 between control and test intervention
Blood pressure | Week 12
  Difference at week 12 between control and test intervention
LDL Cholesterol | week 12
  Difference at week 12 between control and test intervention
Triglycerides | week 12
  Difference at week 12 between control and test intervention
HDL-cholesterol | week 12
  Difference at week 12 between control and test intervention
fasting glucose | week 12
  Difference at week 12 between control and test intervention
fasting insulin | week 12
  Difference at week 12 between control and test intervention

OTHER OUTCOMES:
AST | Week 12
  Difference at week 12 between control and test intervention
creatinine | Week 12
  Difference at week 12 between control and test intervention
Clotting factors | Week 12
  Difference at week 12 between control and test intervention
Subjective symptoms | week 12
  VAS scale, Difference at week 12 between control and test intervention
Dietary change | week 12
  3 day dietary record, difference at week 12 between control and test intervention
ALT | week 12
  Difference at week 12 between control and test intervention

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Vuksan, PhD, Principal Investigator — Unity Health Toronto
Locations (1):
- Clinical Risk Factor and Modification Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jenkins AL, Morgan LM, Bishop J, Jovanovski E, Jenkins DJA, Vuksan V. Co-administration of a konjac-based fibre blend and American ginseng (Panax quinquefolius L.) on glycaemic control and serum lipids in type 2 diabetes: a randomized controlled, cross-over clinical trial. Eur J Nutr. 2018 Sep;57(6):2217-2225. doi: 10.1007/s00394-017-1496-x. Epub 2017 Jul 7. PMID 28687934